CLINICAL TRIAL: NCT02917109
Title: LearningRx Cognitive Training for ADHD: A Multiple Baseline Study Across Cases
Brief Title: LearningRx Cognitive Training for ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gibson Institute of Cognitive Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GICR-0916-A
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LearningRx cognitive training (Experimental): The intervention is a 60-hour, clinician-delivered cognitive training program.
  Interventions: Behavioral: LearningRx cognitive training

INTERVENTIONS:
Behavioral: LearningRx cognitive training — A clinician will deliver three 90-minute cognitive training sessions per week for 14 weeks. There are 16 different categories of leveled training procedures sequenced in intensity and difficulty for a total of 530 training tasks.

SUMMARY:
The purpose of this investigation is to conduct a series of case studies on the impact of LearningRx cognitive training on cognitive skills, brain structure, and daily functioning for participants with ADHD.

DETAILED DESCRIPTION:
Using a multiple baseline design across cases with start point randomization, the proposed study will examine the outcomes from LearningRx one-on-one cognitive training across domains on standardized measures used to monitor treatment effectiveness for ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-22 previously diagnosed with ADHD
* High school students or college students with a prior diagnosis of ADHD living in the greater Colorado Springs area

Exclusion Criteria:

* No braces, metal implants, or claustrophobia that would contraindicate magnetic resonance imaging

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Evidence of overall cognitive function improvement | within 14 days after completing the intervention
  Confirmed by change in pretest to post-test scores on the Woodcock Johnson IV - Tests of Cognitive Abilities

SECONDARY OUTCOMES:
Evidence of change in brain activity | within 30 days after completing the intervention
  As confirmed by pretest to post-test changes in electrical activity measured by qEEG
Evidence of reduction in ADHD symptoms | within 14 days after completing the intervention
  As confirmed by pretest to post-test changes on the ADHD Rating Scale
Evidence of change in brain structure | within 30 days after completing the intervention
  Confirmed by change in pretest to post-test neuroimaging using MRI
Evidence of improvement in visual or auditory attention | with 14 days after completing the intervention
  Confirmed by change in pretest to post-test scores on the Conners Continous Performance Test (CPT-3) and Auditory Attention Test (CATA)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Ledbetter, PhD, Principal Investigator — Gibson Institute of Cognitive Research; Amy L Moore, PhD, Study Director — Gibson Institute of Cognitive Research
Locations (1):
- Gibson Institute of Cognitive Research, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Will add to Harvard Dataverse